CLINICAL TRIAL: NCT06744959
Title: Reliability of Thoracic Trauma Severity Scores in Predicting Outcomes Among Chest Trauma Patients in Low-Resource Settings: A Prospective Cohort Study From Iraq
Brief Title: Thorax Trauma Severity Score in Chest Trauma: A Study in Iraq
Acronym: TTSS-Iraq
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241212B
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chest Trauma
Keywords: TTSS; Chest; Trauma
MeSH Terms: conditions — Thoracic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective observational study aims to evaluate the predictive utility of the Thorax Trauma Severity Score (TTSS) in determining morbidity and mortality in patients presenting with chest trauma at a tertiary hospital in Iraq. The primary objectives of the study are:

To assess the accuracy of TTSS in predicting mortality and critical outcomes such as ICU admission and the need for advanced interventions.

To evaluate the utility of TTSS in stratifying patients based on injury severity in a resource-constrained setting.

To identify demographic and clinical factors influencing the predictive performance of TTSS.

Participants will:

Be assessed using the TTSS upon arrival at the emergency department to establish risk stratification.

Provide demographic and clinical data, including age, gender, mechanism of injury, comorbidities, and length of hospital stay, for analyzing associations with clinical outcomes.

DETAILED DESCRIPTION:
Chest trauma encompasses a wide range of injuries from small rib fractures to potentially fatal thoracic organ injury, making it a major problem in emergency medicine and trauma care. Common causes of chest trauma include motor vehicle collisions (MVCs), falls, and attacks. After head trauma and abdominal damage, chest trauma is the third most prevalent cause of death for patients with polytrauma and the second most common unintended traumatic injury. Death rates from chest trauma are the highest; in some studies, they can reach 60%. Chest trauma is responsible for 25% of mortality in patients with severe trauma. The main causes of death in these situations are frequently ascribed to hypoxia, severe bleeding, or postponed surgery. As such, prompt diagnosis and careful evaluation of the extent of chest damage are essential for enhancing patient outcomes and reducing morbidity and death.

Correct treatment of thoracic trauma, from anticipating the need for urgent care to addressing potential sequelae, depends on an early and precise assessment of the severity level. The requirement for a precise scale in the assessment of thoracic trauma is highlighted by the fact that no scale now in use can accomplish this. Although frequently used, scales like the Trauma Injury Severity Score (TRISS) and the Injury Severity Score (ISS) are global poly-trauma measures that understate localized thoracic damage. The Lung Injury Scale and the Abbreviated Injury Scale (AIStorax) are two other thoracic measures that only use anatomical results. The presence of three or more rib fractures, especially a fracture of the first rib, has traditionally been thought to be related with increased severity. It is currently unclear how factors like age, the mechanism, and the extent of the injury relate to the emergence of pulmonary problems.

Both anatomical and functional criteria were included in the Thorax Trauma Severity Score (TTSS), which was described by Pape et al. in 2000. Using characteristics accessible during the initial examination, the scale was designed to assist emergency medical evaluation in identifying trauma patients at risk of pulmonary problems. This evaluation could be used in both primary and secondary level hospitals. The ability of this scale to predict death has recently been verified. With a score ranging from 0 to 25 points, the TTSS takes into account five important factors: age, pleural injuries, lung contusions, rib fractures, and the PaO2/FiO2 ratio.

Although the TTSS may be useful, its validity about Iraqi hospitals has not yet been fully assessed. This study attempts to close this gap by evaluating the TTSS's prognostic function in forecasting the outcomes of thoracic trauma at tertiary-level hospitals in Iraq. The study aims to ascertain the efficacy of TTSS in a community context and pinpoint precise cut-off points that could help medical professionals make well-informed choices about patient care and treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* patients above 16 years of age.
* Patients presenting to the emergency department with thoracic trauma.
* Patients or their legal guardians must provide informed consent to participate in the study.

Exclusion Criteria:

* Patients with incomplete clinical data or those discharged before scoring can be performed.
* Pregnant patients (due to specific physiological considerations not accounted for by the scoring system).
* Patients who succumb to their injuries before scoring or baseline data collection.
* chronic respiratory diseases
* malignancy and end-organ failure
* Patients with severe head injury (having extradural, subdural, subarachnoid, or intraparenchymal hemorrhage and skull bone fracture) or those requiring prior neurosurgical intervention
* patients with severe abdominal injury requiring surgical intervention like laparotomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes adult patients aged 16 years and older presenting with chest trauma, including both blunt and penetrating injuries, at the emergency department of a tertiary hospital in Iraq. Participants will be evaluated for injury severity using the Thorax Trauma Severity Score (TTSS), with demographic and clinical data collected to explore outcome predictors. This population represents a diverse cohort reflective of trauma patterns in a resource-limited setting.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy Assessment of Thorax trauma severity score (TTSS) in Predicting In-Hospital Mortality | From admission to hospital discharge or death, up to 30 days
  The total score ranges from 0 to 25, with higher scores indicating more severe injuries, a poorer prognosis, and an increased risk of in-hospital mortality.

SECONDARY OUTCOMES:
Accuracy Assessment of the Thorax Trauma Severity Score (TTSS) in Predicting the Need for ICU Admission | From emergency department admission to ICU admission, hospital discharge, or in-hospital death (up to 30 days).
  The TTSS ranges from 0 to 25, with higher scores reflecting more severe thoracic injuries. This outcome evaluates the score's ability to predict the requirement for ICU admission in trauma patients, with higher TTSS values expected to correlate with increased likelihood of ICU admission.
Accuracy Assessment of the Thorax Trauma Severity Score (TTSS) in Predicting Early Hospital Discharge | From hospital admission to discharge, within 72 hours (early discharge).
  This outcome evaluates the ability of the TTSS (ranging from 0 to 25) to predict early hospital discharge in thoracic trauma patients. Lower TTSS values are hypothesized to be associated with a higher likelihood of early discharge, reflecting less severe injury.
Accuracy Assessment of the Thorax Trauma Severity Score (TTSS) in Predicting the Need for Surgical Intervention | From emergency department admission to surgical intervention, hospital discharge, or in-hospital death (up to 30 days).
  This outcome measures the predictive accuracy of the TTSS range (from 0 to 25) in identifying patients who require surgical management (e.g., thoracotomy, VATS, or chest wall repair) due to thoracic trauma. Higher TTSS values are expected to correlate with an increased likelihood of surgical intervention.
Accuracy Assessment of the Thorax Trauma Severity Score (TTSS) in Predicting In-Hospital Morbidity | From hospital admission to discharge or death, up to 30 days.
  This outcome evaluates the incidence and types of complications (morbidity) experienced by patients with thoracic trauma, as predicted by the TTSS range (from 0 to 25). Higher TTSS values are expected to correlate with increased morbidity, including respiratory complications, infections, prolonged mechanical ventilation, and other trauma-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Luma K Mohammed, Assistant professor, Study Director — Al-Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore EE, Malangoni MA, Cogbill TH, Shackford SR, Champion HR, Jurkovich GJ, McAninch JW, Trafton PG. Organ injury scaling. IV: Thoracic vascular, lung, cardiac, and diaphragm. J Trauma. 1994 Mar;36(3):299-300. No abstract available. PMID 8145307
- [Background] Rating the severity of tissue damage. I. The abbreviated scale. JAMA. 1971 Jan 11;215(2):277-80. doi: 10.1001/jama.1971.03180150059012. No abstract available. PMID 5107365
- [Background] Boyd CR, Tolson MA, Copes WS. Evaluating trauma care: the TRISS method. Trauma Score and the Injury Severity Score. J Trauma. 1987 Apr;27(4):370-8. PMID 3106646
- [Background] Bozorgi F, Mirabi A, Chabra A, Mirabi R, Hosseininejad S-M, Zaheri H. Mechanisms of traumatic injuries in multiple trauma Patients. Int J Med Invest. 2018;7:7-15
- [Background] Khandhar SJ, Johnson SB, Calhoon JH. Overview of thoracic trauma in the United States. Thorac Surg Clin. 2007 Feb;17(1):1-9. doi: 10.1016/j.thorsurg.2007.02.004. PMID 17650692
- [Result] Aukema TS, Beenen LF, Hietbrink F, Leenen LP. Validation of the Thorax Trauma Severity Score for mortality and its value for the development of acute respiratory distress syndrome. Open Access Emerg Med. 2011 Aug 23;3:49-53. doi: 10.2147/OAEM.S22802. eCollection 2011. PMID 27147852
- [Result] Pape HC, Remmers D, Rice J, Ebisch M, Krettek C, Tscherne H. Appraisal of early evaluation of blunt chest trauma: development of a standardized scoring system for initial clinical decision making. J Trauma. 2000 Sep;49(3):496-504. doi: 10.1097/00005373-200009000-00018. PMID 11003329
- [Result] Wutzler S, Wafaisade A, Maegele M, Laurer H, Geiger EV, Walcher F, Barker J, Lefering R, Marzi I; Trauma Registry of DGU. Lung Organ Failure Score (LOFS): probability of severe pulmonary organ failure after multiple injuries including chest trauma. Injury. 2012 Sep;43(9):1507-12. doi: 10.1016/j.injury.2010.12.029. Epub 2011 Jan 21. PMID 21256489
- [Result] Clark GC, Schecter WP, Trunkey DD. Variables affecting outcome in blunt chest trauma: flail chest vs. pulmonary contusion. J Trauma. 1988 Mar;28(3):298-304. doi: 10.1097/00005373-198803000-00004. PMID 3351988
- [Result] Chrysou K, Halat G, Hoksch B, Schmid RA, Kocher GJ. Lessons from a large trauma center: impact of blunt chest trauma in polytrauma patients-still a relevant problem? Scand J Trauma Resusc Emerg Med. 2017 Apr 20;25(1):42. doi: 10.1186/s13049-017-0384-y. PMID 28427480